## From Blueprint to Practice: An Innovative Dynamic 9-Box Grid Improves Exercise Participation and Aerobic Capacity in Graduate Students

September 9, 2024

## Informed consent form for graduate nine grid management

## Dear participants:

Hello! We are inviting you to participate in a management experiment titled "The Impact of the Nine-Grid Performance Management on Graduate Students' Aerobic Capacity and Exercise Behavior". This study aims to explore effective methods and their outcomes for enhancing aerobic capacity and exercise participation among graduate students, thereby improving their physical health. The nine-week management cycle will require participants to complete various tasks according to exercise prescriptions designed by the research team throughout the program.

## Rights and obligations of participants

Voluntary Participation: You have the right to voluntarily decide whether to participate in this trial. Your decision will not affect any of your rights and interests at the school; Withdrawal at Any Time: You may choose to withdraw at any stage of the study without giving reasons. Privacy Protection: Your personal information will be strictly confidential, and test data will be processed anonymously without disclosing your identity.

Your Rights: Your research record will contain a unique code used exclusively by the project team for identification purposes. All data storage devices are password-protected, accessible only to authorized members of the project management team. The results of this study may be published in academic publications, journals, or news reports. Your name and other personally identifiable information will not be used for these purposes. Participation in the informed consent form is voluntary. If you decline to participate for any reason, you are not obligated to sign it.

If you have any questions, confusion or complaints about your participation in this study, or have any questions about your rights, you may contact the contact person below this consent form.

Contact: Chen Lei Tel: 13856217003

Informed consent: I have been informed of the purpose, process and possible risks of this trial. All my questions have been answered satisfactorily. I understand that my participation is voluntary and that I can withdraw at any time without adverse effects. The following signature indicates my voluntary consent to participate in this management.

| Signature of participant: | Date: | vear | month | dax |
|---------------------------|-------|--------|-------|-----|
| Signature of participant | Daic | . ycai | | uay |